CLINICAL TRIAL: NCT06021301
Title: Injectable Platelet-Rich Fibrin and Microneedling For Papillae Reconstruction In Esthetic Zone (A Case Series )
Brief Title: Injectable Platelet-Rich Fibrin and Microneedling For Papillae Reconstruction In Esthetic Zone
Acronym: iPRFandMN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmeen Saleh Tolba, Resident at Faculty of Oral and Dental medicine, Cairo University., Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P E R 3-3-1
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Injectable Platelet Rich Fibrin and Microneedling in Papilla Reconstruction; Interdental Papillae Reconstruction
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: Case Series
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iPRF and Microneedling (Experimental): First, MN will be done in the required area with insulin syringe gauge 30,The interdental papilla will vertically and horizontally measured in mm. By establishing a ratio and proportion, the number of microchannels in the region to be treated will calculated to be 250 microchannels per square cm Then, a venous blood sample will be taken for each patient using a 10-ml injector into i-PRF tube containing no anticoagulant and centrifuged at room temperature for 3 min at 700 rpm (60 g force). The 30-gauge dental injector needles will be used for injection of i-PRF. The needle will be inserted at 45° angle, 2-3-mm apical to the involved papilla and all surrounding areas will receive iPRF. Each involved papilla will be injected with an amount till blanching is visible . This method will be repeated for 4 times at 10 days intervals consecutively.
  Interventions: Other: Platelet-Rich Fibrin and Microneedling

INTERVENTIONS:
Other: Platelet-Rich Fibrin and Microneedling — First, MN will be done in the required area with insulin syringe gauge 30,The interdental papilla will vertically and horizontally measured in mm. By establishing a ratio and proportion, the number of microchannels in the region to be treated will calculated to be 250 microchannels per square cm Then, a venous blood sample will be taken for each patient using a 10-ml injector into i-PRF tube containing no anticoagulant and centrifuged at room temperature for 3 min at 700 rpm (60 g force). The 30-gauge dental injector needles will be used for injection of i-PRF. The needle will be inserted at 45° angle, 2-3-mm apical to the involved papilla and all surrounding areas will receive iPRF. Each involved papilla will be injected with an amount till blanching is visible . This method will be repeated for 4 times at 10 days intervals consecutively.

SUMMARY:
The currently available non-surgical techniques for papillary reconstruction did not provide long term maintenance of papillary regeneration, Surgical techniques are invasive and the results are unpredictable . The study is based upon the positive effects of iPRF upon enhancing wound healing in terms of new collagen formation, angiogenesis and increasing keratinized tissue phenotype . iPRF exhibited comparable effects to subepithelial connective tissue graft in papillary reconstruction . The effect of microneedling on the tissue responds as if experiencing tissue trauma and the body's own collagen production is induced to preserve tissue integrity . Growth factors are released immediately after injury, inducing the proliferation of new cells, and fibroblasts are transformed into collagen and elastin fibres from day 5 up to week 8 .

DETAILED DESCRIPTION:
The patients diagnosed with black triangles according to Norland classification system for loss of papillary height will be selected. Each patient will receive a proper knowledge of the study protocols along with full-mouth scaling and root planing (SRP) using ultrasonic and hand instruments and will be given personalized oral hygiene instructions. After oral prophylaxis and baseline measurements of insufficient interdental papilla the treatment will be MN and iPRF. First, MN will be done in the required area with insulin syringe gauge 30,The interdental papilla will vertically and horizontally measured in mm. By establishing a ratio and proportion, the number of microchannels in the region to be treated will calculated to be 250 microchannels per square cm. Then, a venous blood sample will be taken for each patient using a 10-ml injector into i-PRF tube containing no anticoagulant and centrifuged at room temperature for 3 min at 700 rpm (60 g force). The 30-gauge dental injector needles will be used for injection of i-PRF. The needle will be inserted at 45° angle, 2-3-mm apical to the involved papilla and all surrounding areas will receive iPRF. Each involved papilla will be injected with an amount till blanching is visible . This method will be repeated for 4 times at 10 days intervals consecutively. The final clinical photographs and measurements will recorded 3 and 6 months of last dose administered . After the intervention, patients will receive oral hygiene instructions that include the roll technique when brushing without the use of floss and toothpick during the study period to minimize trauma to the treated site .

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking patients aged above 18 years.
* At least one site with interdental papilla recession in the anterior region of the maxillary or mandibular jaws.
* The distance from the contact point to alveolar bone is crest < 7 mm.
* Class I or Class II papillary recession, according to Nordland and Tarnow's classification systems (Nordland et al., 1998).
* No active periodontal diseases and good oral hygiene.

Exclusion Criteria:

* Patients were excluded from the study if they have:
* Spacing or crowding between the teeth to be treated
* Abnormal tooth shape
* Systemic diseases such as diabetes mellitus, hypertension or conditions that alter the outcome of periodontal therapy.
* In addition, patients will be excluded if they are Pregnant and lactating women.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Papillary height | at 3,6 months
  using UNC probe from papillary tip till incisal edge.

CONTACTS AND LOCATIONS:
Overall Officials: yasmeen tolba, Resident, Principal Investigator — department of periodontology ,cairo university
Locations (1):
- Faculty of Dentistry ,Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No